CLINICAL TRIAL: NCT03192436
Title: Electrophysiological Source Imaging Guided Transcranial Focused Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Dr. Bin He, Professor, University of Minnesota
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY2017_00000426
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Ultrasound (Active Comparator): The subjects will receive real ultrasound intervention.
  Interventions: Device: Ultrasound
- Sham Ultrasound (Sham Comparator): The subjects will receive sham ultrasound intervention.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Low-intensity (Ispta < 720 mW/cm2, Isppa < 190 W/cm2) transcranial focused ultrasound

SUMMARY:
Neuromodulation is a fast growing field that offers a wide range of applications for both understanding and treating the brain. Future research for non-invasive neuromodulation will need to elucidate the optimal frequency, duration, and intensity of stimulation for a variety of technologies and diseases. Closed loop stimulation is thus a promising research area that allows for responsive stimulation and real time symptom management. Our project is proposed to develop and test a novel noninvasive neuromodulation integrating transcranial focused ultrasound stimulation (tFUS) with electrophysiological source imaging (ESI-tFUS) to allow evidence-based neuromodulation for brain research and the management of brain conditions. Despite the recent developments and attention surrounding tFUS, relatively little is known about the mechanisms and optimal parameters of this stimulation technology. The addition of ESI neuroimaging, aimed at providing biomarkers to assess the effects of tFUS neuromodulation, could provide crucial necessary information regarding the neural response to the applied stimulation in real-time. In order for tFUS to be further developed and transformed into a robust neuromodulation technology, an integrated electrophysiological source-imaging-guided tFUS system to allow for individualized and responsive stimulation is needed.

The purpose of this study is to develop and evaluate the proposed ESI-tFUS in human subjects using motor and somatosensory paradigms.

DETAILED DESCRIPTION:
In this protocol, the following hypothesis will be tested; the electroencephalography (EEG) and transcranial focused ultrasound (tFUS) will be used to quantify and optimize stimulation effects. We will test the hypothesis that tFUS can induce regional brain activity and use EEG to localize and image the brain electrical activity as induced by TFUS stimulation. Subjects will be recruited for MRI scan and then undergo motor and/or sensory tasks, and during these tasks, subjects will receive tFUS and concurrently be monitored by EEG. This tFUS-EEG study is aimed at exploring effects of tFUS and the use of EEG in providing electrophysiological responses to brain activation following tFUS stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy volunteers.
* Age 18-64.
* Willing and able to provide written consent.
* Able to communicate in the English language.

Exclusion Criteria:

Subjects having any of the following conditions will be excluded from this study:

* Evidence of a current significant medical illness or psychiatric or central or peripheral neurologic disorder
* History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services
* Personal or family history of seizure
* Any history of stroke/transient ischemic attack (TIA)
* Taking any medications that are known to decrease the threshold for seizure
* Pregnancy
* Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully considered by the PI
* Failure to follow laboratory or study procedures

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Closed-loop control of ultrasound neuromodulation as assessed by EEG source imaging | up to 2 years
  The primary study outcome is a closed-loop control algorithm to control the parameters in administrating the tFUS. The outcome data of the study will include the MRI data, EEG data, tFUS location and timing data, perceptual (subject reported) effects of tFUS and/or pins, and any reported adverse events. Analysis of the EEG data will be conducted using EEG analysis software, and the customized software to be developed at the PI's lab. The EEG data will also be correlated with tFUS application. The output of our data analysis process will be in the form of quantitative spatial estimation of tFUS activation in the brain using EEG source reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, Ph.D., Principal Investigator — Carnegie Mellon University
Locations (1):
- Department of Biomedical Engineering, Carnegie Mellon University, Pittsburgh, Pennsylvania, United States